CLINICAL TRIAL: NCT04143074
Title: "Population Activities in the Field of Prevention, Early Identification and Treatment of Overweight and Obesity in Gdansk Children and Youth Population"
Brief Title: Community Based Obesity Prevention and Treatment Programme "6-10-14 for Health"
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Michał Brzeziński (Other)
Responsible Party: Sponsor-Investigator, Michał Brzeziński, Assistant Professor, Primary Investigator, University Clinical Centre, Gdansk
Organization: University Clinical Centre, Gdansk (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NKBBN/228/2012; NKBBN/228/2012 (Other: Independent Bioethics Commission for Research)
Record Dates: First submitted 2019-10-24; First posted 2019-10-29 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Obesity; Obesity, Childhood; Health Program; Body Weight Changes
MeSH Terms: conditions — Obesity; Pediatric Obesity; Body Weight Changes

STUDY DESIGN:
Intervention Model Description: single multidisciplinary intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention (Other): multidisciplinary intervention arm - behavioral intervention by physician, dietician, psychologist and physical activity trainer
  Interventions: Behavioral: multidisciplinary behavioral intervention

INTERVENTIONS:
Behavioral: multidisciplinary behavioral intervention — behavioral intervention - 4 visits with each of the specialist team (pediatrician, dietician, psychologist, physical activity specialist), (4 visits x 4 specialists). Each specialist ap. 30 min time. Wisits in 0-3m-6m-12m time frame. Visits focused on behavioral intervention - motivation for change and basic tools (dietician, physical activity specialist, psychologist) to implement change in nutrition and physical activity based on individual reediness for change (based on Prochaska model).

SUMMARY:
"6-10-14 for Health" is an integrated weight-loss intervention programme for obese children from Gdansk municipality. Both participants of the programme and their family members are offered a 12-month integrated intervention, including medical, dietetic and psychological counselling, as well as educational workshops for parents.

DETAILED DESCRIPTION:
"6-10-14 for Health" is an integrated weight-loss intervention programme for obese children from Gdansk municipality. Both participants of the programme and their family members are offered a 12-month integrated intervention, including medical, dietetic and psychological counselling, as well as educational workshops for parents.

The programme, financed by the municipality of Gdansk, is devided in three phases:

1. Screening - all children aged 6, 9-11, 14 years of age from the City of Gdansk are being screened yearly. All children attending primary and grammar schools in Gdansk are subjected to a screening. The population size is between 9.000-10.000 children yearly.

   All children have anthropometric measurements (body mass, body height, waist circumference), blood pressure, cardiorespiratory fitness.

   Anthropometry: Body weight and body height are determined with a digital scale (Mensor WE150, Poland), with the child wearing an underwear and standing barefoot. Body height is measured to the nearest 0.001 m, and body weight to the nearest 0.1 kg. The scale is calibrated every day. Waist and hip circumferences are measured on a horizontal plane by an Ergonomic Circumference Measuring Tape (model 201; Seca GmbH & Co, KG, Hamburg, Germany).

   Blood pressure measurement: Arterial blood pressure is determined oscillometrically (Omron) on the left arm, with a cuff of an adequate size placed at the level of the heart, in the child seated with uncrossed legs, following at least a 5-min rest in the seated position. The width of the inflatable cuff corresponds to at least 40% of arm circumference. Three separate measurements of blood pressure are taken and averaged.

   Kasch pulse recovery step test: The participants are subjected to a 3-minute Kasch pulse recovery (KPR) step test. The test consists of climbing a 0.305 m step at a rate of 24 steps-up/-down per minute. The rate of climbing is defined by a metronome set at 96 beats (signals) per minute. Heart rate (HR) is monitored continuously with "Polar" (Finland) electronic analyser for 3 minutes of the exercise (step-test) and during 1 minute and 5 seconds of recovery in a seated position. Only post-exercise HR recorded within one minute, starting 5 seconds after completing the test, is subjected to analysis. All HR characteristics are recorded during restitution in a seated position (subjects are instructed to sit still, breath normally and not involve in a conversation). An arithmetic mean calculated from these values (HRmean post-ex) is subjected to further analyses.
2. Intervention - Participants whose anthropometric parameters correspond to overweight (BMI between the 85th and 95th percentile) or obesity (BMI > =95th percentile), according to the percentile charts developed within the framework of the OLAF project, for Poland were qualified to a complex educational and medical intervention for children at increased risk of civilization-related disorders.

Weight- loss intervention programme:

* Dietetic consultation - analysis of nutritional behaviours and dietary habits, selection of appropriate diet. Dietetic consultation takes place at enrolment and 3, 6 and 12 months thereafter.
* Psychological consultation - reinforcement of changes in health behaviours of the child and his/her parents.
* Consultation with a physical education specialist - defining optimal level of physical activity, adjusted to the subject's body weight, abilities and preferences, development of a training programme with increasing intensity and volume of physical activity.

Measurements:

Anthropometry: Body weight and body height are determined with a digital scale (Mensor WE150, Poland), with the child wearing an underwear and standing barefoot. Body height is measured to the nearest 0.001 m, and body weight to the nearest 0.1 kg. The scale is calibrated every day. Waist and hip circumferences are measured on a horizontal plane by an Ergonomic Circumference Measuring Tape (model 201; Seca GmbH & Co, KG, Hamburg, Germany).

Blood pressure measurement: Arterial blood pressure is determined oscillometrically (Omron) on the left arm, with a cuff of an adequate size placed at the level of the heart, in the child seated with uncrossed legs, following at least a 5-min rest in the seated position. The width of the inflatable cuff corresponds to at least 40% of arm circumference. Three separate measurements of blood pressure are taken and averaged [42].

Kasch pulse recovery step test: The participants are subjected to a 3-minute Kasch pulse recovery (KPR) step test [43,44]. The test consists of climbing a 0.305 m step at a rate of 24 steps-up/-down per minute. The rate of climbing is defined by a metronome set at 96 beats (signals) per minute. Heart rate (HR) is monitored continuously with "Polar" (Finland) electronic analyser for 3 minutes of the exercise (step-test) and during 1 minute and 5 seconds of recovery in a seated position. Only post-exercise HR recorded within one minute, starting 5 seconds after completing the test, is subjected to analysis. All HR characteristics are recorded during restitution in a seated position (subjects are instructed to sit still, breath normally and not involve in a conversation). An arithmetic mean calculated from these values (HRmean post-ex) is subjected to further analyses.

Dietetic assessment: Dietary records from three consecutive days (2 weekdays + 1 day of a weekend), collected prior to enrolment and at the end of the intervention are analysed, and dietary intakes of calcium and vitamin D are calculated with Dieta 5.0 software (Institute of Food and Nutrition, Warsaw).

Pubertal status is determined on based on the results of physical examination and expressed using the Tanner stage.

DXA: Total body bone mineral content (TBBMC), total body bone mineral density (TBBMD), lean body mass (LBM), fat mass (FT) (Hologic Discovery Wi)

Laboratory parameters:

Complete blood count Lipid profile determined with an enzymatic method Oral glucose tolerance test (OGTT) with glucose concentration determined with hexokinase method Concentration of insulin determined by means of an immunochemiluminescence assay Concentration of creatinine ALT, TSH, fT4, PTH, Ca, P

Visit 1 (enrolment):

* medical history, physical examination
* interpretation of laboratory findings (tests conducted during screening + concentration of vitamin D),
* anthropometric evaluation and analysis of body composition (bioimpedance method)
* consultation with a dietician, psychologist and specialist in physical activity, and defining detailed protocol of the intervention
* Kasch Pulse Recovery Test

Visit 2 (3 months)

* medical history, physical examination
* anthropometric evaluation and analysis of body composition (bioimpedance method) consultation with a dietician, psychologist and specialist in physical activity, and defining detailed protocol of the intervention. Within a week prior to Visit II - obtaining blood (ca. 5 ml) for laboratory testing (complete blood count, lipid profile, hs-CRP, OGTT, insulin, TSH, fT4).
* consultation with a dietician, psychologist and specialist in physical activity, and defining detailed protocol of the intervention

Visit 3 (6 months)

* medical history, physical examination
* interpretation of laboratory findings
* anthropometric evaluation and analysis of body composition (bioimpedance method)
* consultation with a dietician, psychologist and specialist in physical activity, and defining detailed protocol of the intervention
* obtaining blood for laboratory testing
* termination of active compound/placebo administration

Visit 4 (12 months)

* medical history, physical examination
* anthropometric evaluation and analysis of body composition (bioimpedance method)
* consultation with a dietician, psychologist and specialist in physical activity, and defining detailed protocol of the intervention

The aim of the programme is to reduce baseline body weight of participating children by at least 5% .

ELIGIBILITY:
Inclusion Criteria:

* children living in Gdansk (for screening phase)
* children with BMI above 85 percentile (for intervention phase)
* consent of parent/ caregivers

Exclusion Criteria:

* confirmed congenital or metabolic diseases connected with obesity risk
* lack of consent of parent/ caregivers

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 6000 (Estimated)
Dates: Start 2011-04-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
body mass change | 12 months from begining of intervention
  Number (percentage) of participants with change of: body mass of 5% or centiles of BMI by 5 percentile points or z-score BMI change by 0,25

SECONDARY OUTCOMES:
body fat reduction | 12 months from begining of intervention
  Number (percentage) of participants with change of body fat by at least 5%

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinical Center, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: Undecided
anyone contacting the programme with be assessed and data will be given to researchers/public authorities

REFERENCES:
- See also: protocol abd primary results — https://doi.org/10.1016/j.appet.2014.01.029